CLINICAL TRIAL: NCT02059304
Title: Can Cervical Length Measurement With Embryo Transfer Catheter Predict Preterm Deliveries in ICSI Patients?
Brief Title: Prediction of Preterm Deliveries by Cervical Length Measurement With Embryo Transfer Catheter in ICSI Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Turgut Aydın, Specialist, Gynecology and Obstetrics, Acibadem University
Purpose: Screening
Other Study IDs: CLM PrDelivery Study
Record Dates: First submitted 2014-02-07; First posted 2014-02-11 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Preterm Delivery
Keywords: cervical length; prediction of preterm delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preterm Delivery (Other): Preterm Delivery: Births before the completion of 37 weeks' of gestation.
  Interventions: Device: Measurement of cervical length with embryo transfer catheter
- Term Delivery (Other): Term Delivery: Births after the completion of 37 weeks' of gestation.
  Interventions: Device: Measurement of cervical length with embryo transfer catheter

INTERVENTIONS:
Device: Measurement of cervical length with embryo transfer catheter

SUMMARY:
The aim of this study is to examine the potential value of cervical length (CL) measurement with embryo transfer catheter in the prediction of spontaneous preterm deliveries in intracytoplasmic sperm injection (ICSI) cycles.

Preterm birth is the leading cause of perinatal death and handicap in children. It is clear that ICSI pregnancies are at high risk groupfor preterm delivery (PTD). In singletons there is an estimated two-fold increased risk following ICSI.

CL measurement with ultrasound in mid-trimester (22-24 weeks) is the best method for the prediction of PTD: The shorter the CL, the higher risk of PTD. Recent evidence suggests that at first trimester (11-13 weeks), the risk for PTD is inversely related to CL. It has been shown that the measurement of CL on pregnancy is an effective method for identification of the group at high risk for PTD.

In embryo transfer, catheter is placed the through cervical canal. The method we will use in this study, CL measurement with transfer catheter, will give more precise results than measurement with ultrasound.

No study has been performed to evaluate the prediction of PTD by analyzing measurements of CL, preconceptionally. Our study will be the first in this topic.

There is a certain disadvantage of measuring CL during pregnancy: The effectiveness of prophylactic administrations (progesterone, cervical cerclage etc.) may be inversely related to the gestation at which treatment is initiated. If we know the risk of PTD before gestation, single embryo transfer will be preferred to avoid from multiple pregnancies that also increase the relative risk of PTD, in ICSI pregnancies.

DETAILED DESCRIPTION:
Cervical length measurement protocol: The physician inserted a sterile Collin vaginal speculum; the cervix was exposed and gently cleaned with sterile gauze pads. Cervical mucus was gently removed with a syringe if abundant. A nurse concomitantly performed transabdominal ultrasound scan. Estimated cervical length is determined before transfer procedure. The Sure View Wallace Embryo Replacement Catheter (No. CE118; Smith Medical, Hythe, Kent, UK). There are marked lines on the surface of catheter that show distances to half centimeters. The catheter has a sliding guide fixed at external cervical os. Correct position of the catheter is replaced guide on external os, and guide's endpoint is on internal cervical os. In relation to the internal os was verified on the scan. If required, re-fixation of sliding guide to external os will also be performed. After loading embryos, the length between the guide and the end of catheter will be noted.

Data collection protocol: We will obtain data on pregnancy outcome from the hospital computerized records or the records from family practitioners of the women. We will record birth weeks as major outcome. The obstetric records of all patients will be examined to determine whether any exclusion criteria are present.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women resulting from ICSI treatment at assisted reproduction center, Acibadem Kayseri Hospital, Turkey.

Exclusion Criteria:

* missing outcome data, multiple pregnancies, miscarriages during the first trimester, cigarette smoking, PTD history, progesterone use after 12 weeks, cerclage performed, termination (iatrogenic delivery) and PTDs due to preeclampsia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2012-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Delivery week | Due to the pregnancy period ( maximum 9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Turgut Aydin, Principal Investigator — Acıbadem Kayseri Hospital
Locations (1):
- Acıbadem Kayseri Hospital, Kayseri, Turkey (Türkiye)